CLINICAL TRIAL: NCT03468803
Title: Influence of Open and Laparoscopic Abdominal Surgery Involving the Intestinal Tract on Serum 1,3-ß-D-Glucan (BDG) Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Barmherzige Brueder Marschallgasse / Graz (Unknown)
Responsible Party: Principal Investigator, Robert Krause, MD, Univ.Prof.Dr., Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 30-043 ex 17/18
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Invasive Candidiases
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beta D Glucan (BDG) in surgery (Experimental): Serial Beta D Glucan measurements in each patients before, during, and after surgery
  Interventions: Diagnostic Test: Beta D Glucan test

INTERVENTIONS:
Diagnostic Test: Beta D Glucan test — Measurement of BDG before, during and after surgery

SUMMARY:
Candida species are both known to colonize physiologically mucosal surfaces in the human body without causing signs or symptoms of infection and to cause a wide variety of diseases, including mucocutaneous infections and potentially fatal invasive infections of the bloodstream or organs. Throughout the past decades, invasive fungal infections (IFIs) are of increasing importance even in non-neutropenic patients who are in need of treatment in intensive care units (ICU) or have undergone major surgeries. Several factors like parenteral nutrition, central venous catheters, broad spectrum antibiotics admission, disturbance of gastrointestinal mucosa integrity have been associated with an increased incidence of IFIs. Positive testing for 1,3-ß-D-Glucan (BDG) in serum is widely used to assess invasive fungal infections. It detects circulating BDG, which is part of the fungal cell wall of clinical relevant fungi such as Candida spp. and Aspergillus spp..

The issue of BDG kinetics after intestinal mucosal damage (e.g. mucositis or gut surgery) is poorly understood. Intestinal mucosal damage is characterized by a loss of integrity of the intestinal mucosal barrier and increasing translocations of bacterial and/or fungal commensals of the gastrointestinal tract.

In abdominal surgery a key concern in serum BDG kinetics is the potential introduction of BDG from surgical sponges and gauze or mucosal damage due to surgical damage of the mucosal integrity. Compared to open abdominal surgery in laparoscopic abdominal surgery sponges and gauze are rarely used. As life-threatening intraabdominal candidiasis occurs in 30 to 40% of high-risk abdominal surgical intensive care unit (ICU) patients it is of utmost importance to obtain reliable BDG values for diagnosis or exclusion of invasive candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Elective open abdominal surgery involving the small and/or large colon and with surgical sectioning of intestinal mucosa
* Signed informed consent

Exclusion Criteria:

* Ongoing antifungal therapy for treatment of active fungal infection or antifungal therapy within 4 weeks prior to inclusion
* Antibiotic therapy other than optional single shot surgical prophylaxis as clinically indicated
* Ongoing Enterococcus sp. bacteremia or treatment of Enterococcus sp. bacteremia within 4 weeks prior to inclusion
* Clinical or radiological or laboratory evidence of current infectious disease (i.e. temperature >38°C, elevated C-reactive protein (CRP) >5mg/dl, leukocytosis >11400/μl, elevated neutrophiles >78%) as assessed by the treating physician
* Immunoglobulin, blood or blood products (i.e. thrombocytes, fresh frozen plasma) administration within 4 weeks prior to inclusion
* Abdominal surgery (laparoscopic or open) or other major surgeries (e.g. aortocoronary bypass) within 4 weeks prior to inclusion
* Subsequent invasive candidiasis (defined according to proposed European Organization for Research and Treatment of Cancer Mycoses study group [EORTC/MSG] definitions of fungal infections in ICU) or other complicating infectious disease after surgery within the 5 day observation time frame

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Levels of Beta D Glucan after surgery | after surgery up to day 5
  Measurement of Beta D Glucan after surgery in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Stmk, Austria